CLINICAL TRIAL: NCT05035914
Title: Phase Ib / II Study of Anlotinib Combined With mXELIRI as Second-line Treatment of Advanced Colorectal Cancer
Brief Title: Anlotinib Combined With mXELIRI as Second-line Treatment of Advanced Colorectal Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangzhou University of Traditional Chinese Medicine (Other)
Collaborators: Guangdong Provincial Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Guangzhouucm
Record Dates: First submitted 2021-09-03; First posted 2021-09-05 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Advanced Colorectal Cancer
Keywords: advanced colorectal cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: anlotinib+mXELIRI (Experimental): Dose-escalation phase:
  A: anlotinib 8 mg, po, qd, d1-14; iritecan 180-200mg/m2, iv, d1;capecitabine 800mg/m2, po, bid, d1-14; every 3 weeks as a cycle;
  B: anlotinib 10 mg, po, qd, d1-14; iritecan 180-200mg/m2, iv, d1;capecitabine 800mg/m2, po, bid, d1-14; every 3 weeks as a cycle;
  C: anlotinib 12 mg, po, qd, d1-14; iritecan 180-200mg/m2, iv, d1;capecitabine 800mg/m2, po, bid, d1-14; every 3 weeks as a cycle;
  Dose-expansion phase:
  anlotinib RP2D, po, qd, d1-14; iritecan 180-200mg/m2, iv, d1;capecitabine 800mg/m2, po, bid, d1-14; every 3 weeks as a cycle;
  Interventions: Drug: Anlotinib Hydrochloride

INTERVENTIONS:
Drug: Anlotinib Hydrochloride — Anlotinib Hydrochloride is a capsule in the form of 8 mg ,10 mg and 12 mg, orally, once daily, 2 weeks on/1 week off.

SUMMARY:
1. Determine the maximum tolerable dose (MTD) and / or phase II recommended dose (RP2D) of the allotinib combined mXELIRI protocol.
2. To evaluate the safety and tolerance of the combination of anlotinib and mXELIRI in the second-line treatment of patients with advanced colorectal cancer

DETAILED DESCRIPTION:
This study consists of two phases, the dose-escalation phase, and the expansion phase. 9-12 patients with advanced colorectal cancer will be included in the dose escalation study. Patients who met the inclusion criteria would be treated with anlotinib QD for 2 weeks, and then stopped for 1 week, combined with mXELIRI. Every 21 days was a treatment cycle. Safety information was collected until the disease progression or intolerable toxicity, so as to determine the MTD and / or RP2D of anlotinib combined with irinotecan in patients with advanced colorectal cancer. The study adopted the traditional 3+3 design .

The primary outcome in dose-expansion phase was objective response rate(ORR).

ELIGIBILITY:
Inclusion Criteria:

* ECOG performance status (PS) 0-1
* The expected survival time is not less than 12 weeks
* Patients with stage IV colorectal cancer confirmed by pathology or imaging have measurable lesions (according to RECIST 1.1, the long diameter of tumor lesions on CT scan is greater than or equal to 10 mm, the short diameter of lymph node lesions on CT scan is greater than or equal to 15 mm, and the measurable lesions have not received radiotherapy, freezing and other local treatment);
* First line patients with advanced or intolerant colorectal cancer treated with bevacizumab combined with oxaliplatin (FOLFOX or capeox, etc.);
* The function of main organs was normal (in accordance with the chemotherapy standard);
* Women of childbearing age must have taken reliable contraceptive measures or conducted pregnancy test (serum or urine) within 7 days before enrollment, and the result is negative, and they are willing to use appropriate contraceptive methods during the test period and 8 weeks after the last administration of the test drug. For men, it is necessary to agree to use appropriate contraceptive methods or surgical sterilization during the trial period and 8 weeks after the last administration of the trial drug;
* The subjects volunteered to join the study and signed informed consent, with good compliance and follow-up.

Exclusion Criteria:

* The histological type was mucinous adenocarcinoma or ovarian implant metastasis;
* First line patients with irinotecan treatment;
* Patients who had been treated with anlotinib hydrochloride capsules in the past;
* Symptomatic brain metastases (patients with stable symptoms and completed treatment 21 days before enrollment can be enrolled, but no cerebral hemorrhage symptoms should be confirmed by brain MRI, CT or venography evaluation);
* Patients with hypertension who could not be well controlled by single antihypertensive drug treatment (systolic blood pressure ≥ 150 mmHg, diastolic blood pressure ≥ 100 mmHg); Or use two or more antihypertensive drugs to control blood pressure
* The patient also had more than 1 degree of adverse reactions (except hair loss, neurotoxicity more than 2 degrees) which could not be alleviated due to previous treatment;
* They have the following cardiovascular diseases: myocardial ischemia or myocardial infarction above grade II, poorly controlled arrhythmias (including QTc interval ≥ 450 ms for male and ≥ 470 MS for female); According to NYHA criteria, grade Ⅲ - Ⅳ cardiac insufficiency, or left ventricular ejection fraction (LVEF) < 50% by echocardiography;
* Abnormal coagulation function (INR > 1.5 or PT > ULN + 4 seconds or APTT > 1.5 ULN), bleeding tendency or receiving thrombolysis or anticoagulation therapy;
* There were significant clinical bleeding symptoms or clear bleeding tendency in the first 3 months, such as gastrointestinal bleeding, hemorrhagic hemorrhoids, hemorrhagic gastric ulcer, baseline fecal occult blood + + or above, or vasculitis;
* Arteriovenous thrombotic events occurred in the first 12 months, such as cerebrovascular accident (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), deep venous thrombosis and pulmonary embolism;
* Known hereditary or acquired bleeding and thrombotic tendency (such as hemophilia, coagulation dysfunction, thrombocytopenia, hypersplenism, etc.);
* Wound or fracture that has not been cured for a long time (pathological fracture caused by tumor is not included);
* Patients in the study group had undergone major surgery or severe traumatic injury, fracture or ulcer within 4 weeks;
* There are obvious factors affecting oral drug absorption, such as inability to swallow, chronic diarrhea and intestinal obstruction;
* Abdominal fistula, gastrointestinal perforation or abdominal abscess occurred within 6 months before admission;
* Urine routine showed that urine protein was ≥ + +, and 24-hour urine protein was more than or equal to 1.0 G;
* Serous effusion (including pleural effusion, ascites and pericardial effusion) with clinical symptoms and requiring symptomatic treatment;
* Asymptomatic serous effusion can be included in the group, symptomatic serous effusion after active symptomatic treatment (can not use anticancer drugs for serous effusion treatment), patients who can be included in the group after the judgment of the researchers are allowed to be included in the group.
* Active infections need antimicrobial treatment (for example, the use of antibiotics and antiviral drugs, excluding chronic hepatitis B anti hepatitis B treatment, antifungal treatment).
* There was active hepatitis B (HBV DNA > 2000IU/mL or 104 copy number /mL) or hepatitis C (hepatitis B antibody positive, and HCV RNA was higher than the lower limit of analysis).
* Those who have a history of psychotropic drug abuse and can not give up or have mental disorders;
* Those who participated in clinical trials of other anti-tumor drugs within 4 weeks before enrollment;
* Previous or other untreated malignancies were cured except for basal cell carcinoma, cervical carcinoma in situ and superficial bladder cancer.
* Those who received strong CYP3A4 inhibitor treatment within 7 days before randomization, or those who received strong CYP3A4 inducer treatment within 12 days before participating in the study;
* Pregnant or lactating women; Patients with fertility are unwilling or unable to take effective contraceptive measures;
* The researcher judges other situations that may affect the clinical research and the judgment of research results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2021-07-09 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | Through study completion, up to 24 months
  The main side effects of drugs are the main reasons for limiting the increase of the dose of chemotherapy drugs, which are dose limiting toxicity of chemotherapy drugs
Phase II clinical recommended dose (RP2D) | each 42 days up to intolerance the toxicity or PD
  When the minimum number of patients is included in the dose increasing phase, the recommended dose of phase 2 can be determined accurately and quickly
Objective response rate | Through study completion, up to 24 months
  Objective response rate is defined as the percentage of subjects with evidence of a confirmed complete response (CR) or partial response (PR) as per Response Evaluation Criteria In Solid Tumors (RECIST) Version 1.1.prior to progression or any further therapy.

SECONDARY OUTCOMES:
Progression free survival | From date of enrollment until the date of first documented progression, assessed up to 24 months
  Progress free survival defined as the time from first dose of study treatment until the first date of either objective disease progression or death due to any cause
Overall survival | From date of enrollment until death, assessed up to 24 months
  Overall survival is defined as the time until death due to any cause
Disease control rate | Through study completion, up to 24 months
  Defined as the proportion of patients with a documented complete response, partial response, and stable disease (CR + PR + SD) based on RECIST 1.1
Duration of remission | Through study completion, up to 24 months
  The time from the first time that CR or PR (no matter which one is measured first) is measured to the first time that disease recurrence or progression is truly recorded
Score of quality of Life | From date of enrollment until death, assessed up to 24 months
  The changes of clinical symptoms and objective examination results of tumor patients before and after treatment were observed and scored. According to the requirements of quality of life scale, the scoring results of each field of the scale were recorded in ECRF

CONTACTS AND LOCATIONS:
Overall Officials: Haibo Zhang, Professor, Principal Investigator — Guangdong Provincial Hospital of Traditional Chinese Medicine
Locations (1):
- Guangdong Provincial Hospital of Chinese Medicine, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No